CLINICAL TRIAL: NCT01202357
Title: Community Case Management for Early Psychosis: is Two Year an Optimal Duration? A Randomized Controlled Study
Brief Title: Optimal Duration of Early Intervention for Psychosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: Queen Mary Hospital, Hong Kong (Other); Pamela Youde Nethersole Eastern Hospital (Other); Kwai Chung Hospital (Other)
Responsible Party: Prof. Eric Y. H. Chen, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CM-RCT
Record Dates: First submitted 2010-09-13; First posted 2010-09-15 (Estimated); Last update posted 2010-09-15 (Estimated); Status verified 2010-09

CONDITIONS: Psychotic Disorders
Keywords: Psychotic Disorders; Psychosis
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Case Management (1 year) (Experimental)
  Interventions: Behavioral: Community Case Management
- Standard Care (1 year) (No Intervention)
  Interventions: Behavioral: Community Case Management

INTERVENTIONS:
Behavioral: Community Case Management — Community case management for psychosis by designated key-worker according to specified protocol

SUMMARY:
A total of 160 subjects, who aged 18-35 and had completed the first 2 years of case management in the EASY programme will be randomized in 1:1 ratio into either (1) receiving an additional year of case management, or (2) terminating case management for the next 12 months. The current study aims to investigate whether an additional year of case management in year 3 will confer additional benefits in outcome, in terms of functioning, symptoms, quality of life and health economics.

DETAILED DESCRIPTION:
Psychotic disorders involve disturbances in perceptual, cognitive and motivational processes central to the human life experience, which resulting in long-term and pervasive functional disability. In order to achieve the best possible long-term community outcome of psychotic disorders, early intervention service is set up, focusing on the first few years (the critical period) of the illness.

In Hong Kong, early intervention for psychotic disorder was provided since 2001. The integrated Early Assessment Service for Young people with psychosis (EASY) provide specialized care to early psychosis patients up to age 25. Evaluation of the EASY programme using a matched historical control suggesting that early intervention is a promising approach to promote community care for patients with psychosis.

In the current service, case management for patients will terminate after two years, and the patients will make transition to general psychiatric care afterwards. It is not clear whether the provision of additional case management in the community (e.g., for another year) will significantly enhance outcome further.

The proposed study aims to investigate the effectiveness of providing community based case management for an additional year for patients with psychotic disorders by using a randomized controlled design. The study recruit patients who had completed the first 2 years of case management in the EASY programme and randomized them to receive either an additional year of case management, or to terminate case management for the next 12 months. The hypothesis is that better outcome are found in patients who had 3-year case management compared with those who had only 2 years.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of schizophrenia, schizophreniform disorder, schizoaffective disorder, brief psychotic disorder, psychosis not otherwise specified or delusional disorder
* Received EASY service for 2 years following a first-episode psychosis
* Cantonese-speaking Chinese
* Ability to understand the study and to provide written informed consent

Exclusion Criteria:

* Organic brain disorder
* Known history of intellectual disability
* Drug-induced psychosis

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2010-07; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Functioning (social and occupational) | baseline, 12-month

SECONDARY OUTCOMES:
Symptoms, quality of life and health economics | baseline, 12-month

CONTACTS AND LOCATIONS:
Overall Officials: Eric YH Chen, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, China

REFERENCES:
- [Derived] Chang WC, Kwong VWY, Lau ESK, So HC, Wong CSM, Chan GHK, Jim OTT, Hui CLM, Chan SKW, Lee EHM, Chen EYH. Sustainability of treatment effect of a 3-year early intervention programme for first-episode psychosis. Br J Psychiatry. 2017 Jul;211(1):37-44. doi: 10.1192/bjp.bp.117.198929. Epub 2017 Apr 6. PMID 28385705